CLINICAL TRIAL: NCT00181766
Title: A Pilot Study of Strattera Treatment in Adults With Attention Deficit Hyperactivity Disorder Not Otherwise Specified
Brief Title: Strattera Treatment in Adults With Attention Deficit Hyperactivity Disorder Not Otherwise Specified (ADHD NOS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD; Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-P-002052
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2010-06-23 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: ADHD NOS
Keywords: ADHD NOS; Adults; Strattera (atomoxetine); Open-Label
MeSH Terms: interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Strattera (atomoxetine) (Experimental)
  Interventions: Drug: Strattera (atomoxetine)

INTERVENTIONS:
Drug: Strattera (atomoxetine) — Up to maximum of 1.2mg atomoxetine/kg PO QD, or 120 mg atomoxetine PO QD (whichever is less).
  Other Names: Strattera

SUMMARY:
This is an open-label study with daily doses up to 144 mg/day Strattera (atomoxetine) in the treatment of adults with attention deficit hyperactivity disorder not otherwise specified. The researchers hypothesize ADHD symptomatology in adults with ADHD NOS will be responsive to Strattera treatment and Strattera treatment (in doses of up to 120 mg/day or 1.5 mg/kg/day, whichever is less) in adults with ADHD NOS will be safe and well tolerated.

DETAILED DESCRIPTION:
Strattera (atomoxetine) is a non-stimulant specific norepinephrine reuptake inhibitor recently approved by the Food and Drug Administration for the treatment of child, adolescent and adult patients with ADHD. It is possible Strattera could be a viable alternative treatment for ADHD individuals. The purpose of this study is to assess the effectiveness, safety and tolerability of Strattera in adults with ADHD NOS. If this initial study shows promise, we will follow-up with a randomized clinical trial.

The study includes:

1. use of a six-week design to document the response rate,
2. weekly assessments to document the impact of Strattera NOS on functional capacities,
3. careful assessment of safety and tolerability.

Primary outcomes measure symptom reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients older than 18 and younger than 55 years of age.
2. Subjects with the diagnosis of attention deficit hyperactivity disorder not otherwise specified (ADHD NOS), by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), as manifested in clinical evaluation and confirmed by structured interview. This is operationalized by either:

   1. having currently at least 6/9 current items of either inattention or hyperactivity/impulsivity but < 5 items from either list in childhood; or
   2. having 5 out of 9 current DSM-IV items of inattention and/or hyperactivity/impulsivity, but not having 6 current symptoms in either category. This second category will be included independent of the presence or absence of ADHD symptoms in childhood.
3. Subjects will have a current Clinical Global Impression ADHD score of 4 or higher.
4. Subjects with past history of depression or anxiety disorder (including obsessive compulsive disorder [OCD]) without current disorder for > 3 months as ascertained through structured diagnostic interview and clinical exam will be allowed to participate.
5. Subjects treated for anxiety disorders and depression who are on a stable medication regimen for at least three months, and who have a disorder specific CGI-severity score ≤ 3 (mildly ill) and who have a score on the Hamilton-depression and Hamilton-anxiety rating scale below 15 (mild range) will be included in the study.
6. Subjects with past history of substance use disorders but have been asymptomatic for at least 6 months and have a negative drug screen will be allowed to participate.
7. Subjects receiving non-monoamine oxidase inhibitor (MAOI) antidepressants (e.g., selective serotonin reuptake inhibitors [SSRIs], bupropion, venlafaxine), or benzodiazepines who have been on a stable regimen for > 3 months for any of the conditions listed above.
8. Subjects with mild cases of asthma and allergy will be allowed to participate.
9. Subjects with acid reflux syndrome will be allowed to participate.
10. Subjects with hypercholesterolemia who are on a stable dose of cholesterol-lowering medication will be allowed to participate.

Exclusion Criteria:

1. Any clinically unstable psychiatric conditions including the following: acute psychosis, acute panic, acute OCD, acute mania, acute suicidality, lifetime history of bipolar disorder, acute substance use disorders (alcohol or drugs), sociopathy, criminality.
2. Any metabolic, neurological, hepatic, renal, cardiovascular, hematological, ophthalmic, or endocrine disease.
3. Clinically significant abnormal baseline laboratory values which include the following:

   1. Values larger than 20% above the upper range of the laboratory standard of a basic metabolic screen.
   2. Exclusionary blood pressure parameters will include any values above 140 (systolic) and 90 (diastolic).
   3. Exclusionary electrocardiogram (ECG) parameters will include a QTC > 460 msec, QRS > 120 msec, and PR > 200 msec. Subjects having ECG evidence of ischemia or arrhythmia as reviewed by an independent cardiologist.
4. Mental retardation (intelligence quotient [I.Q.] < 75).
5. Organic brain disorders.
6. Pregnant or nursing females.
7. Subjects with current adequate treatment for ADHD or a history of a previous adequate trial of Strattera.
8. Subjects who have failed to respond to an adequate trial, or who have had tolerability problems on Strattera.
9. Only English-speaking subjects will be allowed into the study for the following reasons:

   1. the assessment instruments are not available and have not been adequately standardized in other languages;
   2. the researchers' clinical trials facility is located in Cambridge and not in the Massachusetts General Hospital (MGH) main campus without the availability of translators;
   3. psychiatric questionnaires and evaluations are taxing and adding the complexity of a translator has the potential to make the patient experience even more exhausting.
10. Prior hypersensitivity to Strattera.
11. MAOI antidepressant use currently or within two weeks of starting study.
12. Urinary retention or bladder dysfunction.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2003-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were from referrals to the Adult ADHD Program at the MGH and through advertisements in the local media. The majority of subjects referred to our program first participate in our general screening protocol entitled, "A Screening Protocol for Adults with Attention Deficit Hyperactivity Disorder" (Protocol # 2002-P-001856).
Groups:
- Strattera (Atomoxetine): Atomoxetine monotherapy up o 1.2 mg/kg/day or 120 mg/day.
Period: Overall Study
Arm/Group | Strattera (Atomoxetine)
Started | 45 (Number of subjects enrolled and treated with Atomoxetine.)
Completed | 33 (Completed the trial.)
Not Completed | 12
Not completed — Lost to Follow-up | 6
Not completed — Adverse Event | 4
Not completed — non-compliance | 2

BASELINE CHARACTERISTICS:
Arm/Group | Strattera (Atomoxetine)
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: ADHD-Clinical Global Impression
Description: The CGI includes Global Severity (1=not ill; 7=extremely ill) and the Global Improvement (1=very much improved; 7=very much worse) Scales. Overall severity and change in severity of ADHD was assessed with the Clinical Global Impression Scale (CGI). Improvement was defined by CGI-I ≤2, much or very much improved, at study endpoint. Results are given as number of subjects who improved according to the CGI-I using the definition above.
Time Frame: 6 Weeks
Population: All analyses were intention to treat (ITT) with the last observation carried forward (LOCF) for subjects who did not complete the full study schedule.
Measure: Number; unit: subjects
Arm/Group | Strattera (Atomoxetine)
Number analyzed (Participants) | 45
subjects | 29

2. Primary Outcome: The Adult AISRS
Description: The Adult AISRS was used to assess each of the 18 individual criteria symptoms (both inattentive and hyperactive) of ADHD in DSMIV on a severity grid (0=not present; 3=severe; minimum score=0; maximum score=54). Results are given as average change (reduction) in AISRS symptoms from baseline to Week 6.
Time Frame: baseline and 6 Weeks
Population: All analyses were intention to treat (ITT) with the last observation carried forward (LOCF) for subjects who did not complete the full study schedule. Baseline and endpoint AISRS scores were compared used paired t-tests. Statistical significance was determined at alpha level 0.05.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Strattera (Atomoxetine)
Number analyzed (Participants) | 45
scores on a scale | -12.1 (8.4)

ADVERSE EVENTS:
Arm/Group | Strattera (Atomoxetine)
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 45/45
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Strattera (Atomoxetine) (N=45)
Dry Mouth (Gastrointestinal disorders) | 26
Gastrointestinal (Gastrointestinal disorders) | 22
Insomnia (General disorders) | 22
Tired/fatigued (General disorders) | 22
Headache (General disorders) | 17
Decreased appetite (Metabolism and nutrition disorders) | 15
Warmth/flushing/sweating (Nervous system disorders) | 13
Colds/allergies/infections (Immune system disorders) | 11
Lightheaded/dizzy (General disorders) | 10
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 9
Tension/jitteriness (Nervous system disorders) | 9
Mood change (Psychiatric disorders) | 7
Sexual function (Reproductive system and breast disorders) | 7
Urinary hesitancy (Renal and urinary disorders) | 6
Neurologic (Nervous system disorders) | 5
Vision/ocular (Eye disorders) | 5
Feeling cold (Nervous system disorders) | 4
Injury (Injury, poisoning and procedural complications) | 4
Muscle twitch/tremor (Musculoskeletal and connective tissue disorders) | 4
Impaired concentration (Nervous system disorders) | 3
Palpitations (Cardiac disorders) | 3
Tingling sensation (Nervous system disorders) | 3
Vivid dreams (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 2
Bad taste (Nervous system disorders) | 2
Chest discomfort (Cardiac disorders) | 2
Skin changes (Skin and subcutaneous tissue disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 1
Paresthesia (Nervous system disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1

LIMITATIONS AND CAVEATS:
* small, open label study
* short exposure to medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No